CLINICAL TRIAL: NCT07212179
Title: Safety and Feasibility of a Self-Learning Bolus Calculator With Simplified Meal Announcement in Adolescents With Type 1 Diabetes Using Automated Insulin Delivery
Acronym: InsuLearn-SMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anas El Fathi (Other)
Responsible Party: Sponsor-Investigator, Anas El Fathi, Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 302850
Record Dates: First submitted 2025-09-29; First posted 2025-10-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes (T1D); Automated Insulin Delivery (AID); Continuous Glucose Monitor (CGM); Diabetes Assistant (DiAs); Carbohydrate Counting (CC); Simplified Meal Announcement (SMA)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- AID + InsuLearn-SMA (Experimental): Participant will use their Automated insulin delivery (AID) system [insulin pump] along with InsuLearn simplified meal announcement bolus calculator
  Interventions: Device: AID + InsuLearn-SMA
- Carbohydrate Counting (Placebo Comparator): Participant will use their Automated insulin delivery (AID) system [insulin pump] and their usual carbohydrate counting bolus calculator
  Interventions: Device: AID + CC

INTERVENTIONS:
Device: AID + InsuLearn-SMA — Automated insulin delivery (AID) system with InsuLearn simplified meal announcement bolus calculator
  Arms: AID + InsuLearn-SMA
Device: AID + CC — Automated insulin delivery (AID) system using usual carbohydrate counting bolus calculator
  Arms: Carbohydrate Counting

SUMMARY:
To evaluate the safety and feasibility of a novel self-learning bolus calculator along with simplified meal announcement (AID+InsuLearn-SMA) in adolescents and young adults with T1D using Automated Insulin Delivery.

DETAILED DESCRIPTION:
Following recruitment and screening, participants will be randomized to one of two sequences during the Hotel Admission: AID+InsuLearn-SMA→AID+CC or AID+CC→AID+InsuLearn-SMA. All participants will be trained on the study equipment, which includes (i) the DiAs smartphone running the Control-IQ algorithm with either the InsuLearn-SMA bolus calculator or the standard carbohydrate counting bolus calculator, and (ii) the Dexcom CGM. All participants will complete 7 days/6 nights run-in At-Home Period using the AID+CC system (Control-IQ with the standard carbohydrate counting bolus calculator). Participants will then undergo a 2-night supervised hotel admission (approximately 48 hours). During this admission, each participant will consume two standardized meals (dinner and breakfast), during which either the InsuLearn-SMA bolus calculator or the standard CC bolus calculator will be used in a randomized order. Two lunches will be offered during the Hotel Admission but not included in the analysis. Following discharge, all participants will complete 7 days/6 nights At-Home Period using the AID+InsuLearn-SMA system before returning the study equipment. The INSPIRE Questionnaire will be administered before and after the Hotel Admission. Additionally, participants will be asked to provide a 2-week CGM data download of their usual care for statistical analysis before randomization and after returning the equipment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥14.0 and ≤21 years old at time of consent
2. HbA1c ≤ 10%.
3. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
4. Having used an insulin pump within the last three months.
5. Currently using insulin for at least six months
6. Willingness to use insulin parameters such as carbohydrate ratio and correction factors consistently on their pump in order to dose insulin for meals or corrections
7. Willingness to switch to a commercially approved insulin (e.g. lispro or aspart or biosimilar approved products) within the study pump as directed by the study team.
8. Has one or more supportive caregivers or companions living with the participant who are knowledgeable about emergency procedures for treatment of severe hypoglycemia and able to contact emergency services and study staff.
9. Acceptable forms of contraception for participants of child-bearing potential include hormonal treatments including IUD, abstinence from heterosexual intercourse, vasectomy in partner, barrier methods (e.g. condom or diaphragm).
10. For females, not currently known to be pregnant or breastfeeding. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
11. Willingness to use the study InsuLearn system (CGM, pump, and phone) during the study period.
12. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial.
13. Access to internet at home and ability to upload data during the study as needed.
14. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol.
15. Participant is proficient in reading and writing English.

Exclusion Criteria:

1. History of diabetic ketoacidosis (DKA) in the 12 months prior to enrollment
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
3. Pregnancy or intent to become pregnant during the trial
4. Currently breastfeeding or planning to breastfeed
5. Currently being treated for a seizure disorder
6. Planned surgery during study duration
7. History of cardiac arrhythmia (except for benign premature atrial contractions and benign premature ventricular contractions which are permitted)
8. Treatment with any non-insulin glucose-lowering agent (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and naturaceuticals)
9. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
10. Participation in another interventional trial at the time of enrollment.
11. Visual impairment/blindness that prevents proper interaction with study equipment
12. Participant who may have a falsely eligible HbA1c due to medical conditions or blood donations.
13. Participants in whom the G6 CGM may be inaccurate due to interference.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
TIR (70-180 mg/dL) | 18 hours
  The primary outcome will be the CGM-measured time in range (TIR, 70-180 mg/dL) during the hotel portion.

SECONDARY OUTCOMES:
TIR (70-180 mg/dL) | 1-week
  The primary outcome will be the CGM-measured time in range (TIR, 70-180 mg/dL) during the at-home period.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Schoelwer, MD, Principal Investigator — University of Virginia School of Medicine
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States